CLINICAL TRIAL: NCT01923259
Title: Single Dose Crossover Comparative Bioavailability Study of Donepezil 23 mg Tablets in Healthy Male and Female Volunteers / Fed State
Brief Title: Bioavailability Study of Donepezil Hydrochloride Tablets 23 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DNI-P0-653
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil Hydrochloride Tablets, 23 mg (Experimental): Donepezil Hydrochloride Tablets, 23 mg of Dr.Reddy's Laboratories Ltd
  Interventions: Drug: Donepezil
- Aricept (Active Comparator): Aricept® 23 mg tablet of Eisai Inc
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil Hydrochloride tablets,23 mg
  Other Names: Aricept

SUMMARY:
To evaluate and compare the relative bioavailability and therefore the bioequivalence of two different formulations of donepezil after a single oral dose administration under fed conditions.

DETAILED DESCRIPTION:
Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover study under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteer
2. Volunteer aged of at least 18 years but not older than 45 years
3. Volunteer with a body mass index (BMI) greater than or equal to 21 and below 30 kg/m2
4. Volunteer with a body weight greater than or equal to 60 kg.
5. Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before day 1 of this study. An ex-smoker is defined as someone who completely stopped smoking for at least 12 months before day 1 of this study.
6. Availability for the entire study period
7. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee.
8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis)
10. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer

Exclusion Criteria

1. Seated pulse rate less than 50 bpm at screening
2. Seated blood pressure below 105/60 mmHg at screening
3. Seated blood pressure below 105/60 mmHg before drug administration
4. Females who are pregnant or are lactating
5. Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study
6. History of significant hypersensitivity to donepezil, piperidine derivatives, scopolamine, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
7. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
8. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
9. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
10. Suicidal tendency, history of or disposition to seizures, state of confusion,clinically relevant psychiatric diseases
11. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS >110 msec and QTc > 440 msec) on the screening ECG or other clinically significant ECG abnormalities.
12. Use of ASA or NSAIDs (or any product containing ASA or NSAIDs) in the previous 7 days before day 1 of this study
13. Use of diphenhydramine in the previous 10 hours before day 1 of this study
14. Known presence of rare hereditary problems of galactose and /or lactose intolerance
15. Known presence of glaucoma or a predisposition to angle-closure glaucoma
16. Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
17. Any clinically significant illness in the previous 28 days before day 1 of this study
18. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
19. Any history of tuberculosis and/or prophylaxis for tuberculosis
20. Positive urine screening of alcohol and/or drugs of abuse
21. Positive results to HIV, HBsAg or anti-HCV tests
22. Females who are pregnant according to a positive serum pregnancy test
23. Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study.
24. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 18, 24, 48 and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada